CLINICAL TRIAL: NCT02028585
Title: Effects of Low-fat Milk Consumption on Metabolic and Atherogenic Biomarkers in Korean Adults With Metabolic Syndrome: a Randomized Controlled Trial
Brief Title: Effects of Low Fat Milk Consumption on Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Food and Drug Safety, Korea (Other Government)
Responsible Party: Principal Investigator, Nan Hee Kim, Prof, Korea University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12162-mfds-118; 12161MFDS118 (Other Grant/Funding Number: Ministry of Food and Drug Safety)
Record Dates: First submitted 2013-12-30; First posted 2014-01-07 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2013-12

CONDITIONS: Metabolic Syndrome
Keywords: low-fat milk; metabolic syndrome; lipid profile; inflammation; oxidative stress; endothelial function
MeSH Terms: conditions — Metabolic Syndrome; Inflammation

ARMS (2):
- Low-fat milk group (Active Comparator): The low-fat milk group was instructed to consume 2 packs of low-fat milk per day (200 mL twice daily) for 6 weeks.
  Interventions: Dietary Supplement: Low-fat milk group
- Control group (No Intervention): Control group maintained their usual diet without low-fat milk supplement.

INTERVENTIONS:
Dietary Supplement: Low-fat milk group
  Arms: Low-fat milk group

SUMMARY:
This study aimed to investigate the effects of low-fat milk consumption on metabolic parameters and biomarkers related to inflammation, oxidative stress, and endothelial function in Korean adults with metabolic syndrome.

DETAILED DESCRIPTION:
A randomized, controlled, parallel, dietary intervention study was designed. Subjects with metabolic syndrome and body mass index ≥23 kg/m2 were randomized to the low-fat milk group, which were instructed to consume 2 packs of low-fat milk per day (200 mL twice daily) for 6 weeks, and the control group was instructed to maintain their habitual diet. Metabolic markers were evaluated at baseline and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were enrolled if their body mass index (BMI) was ≥23 kg/m2 and they met the criteria for metabolic syndrome.

Exclusion Criteria:

* Those who were allergic to milk; those who had a history of digestive disorder; those with a medical history of cardiovascular diseases, including coronary artery diseases, valvular heart diseases, heart failure, or stroke; those who had cancer in the past 5 years; those who were taking hypoglycemic agents for diabetes mellitus; those who had chronic disease such as renal failure or liver cirrhosis; and those with a hemoglobin A1c (HbA1c) level ≥ 7% were excluded from the research. People who had a weight change > 5% of the total weight within the past 3 months, those who had started taking or had changed their dose of anti-hypertensive agents or medications for dyslipidemia within the previous 1 month, those who had a newly diagnosed dyslipidemia requiring drug treatment, those who had taken steroids either orally or by injection within the previous 3 months, those who were pregnant or were expecting to become pregnant; and those who regularly consumed milk in quantities ≥ 200 mL per day at least 3 times a week on average were also excluded.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-04; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
metabolic parameters | 6 weeks
  lipid profiles, body mass index, waist circumference, blood pressure, fasting glucose, insulin, hemoglobin A1c and homeostasis model assessment of insulin resistance
inflammation markers | 6 weeks
  white blood cell count, high-sensitive C-reactive protein, Interleukin-6, adiponectin, serum and urine malondialdehyde, oxidized low-density lipoprotein, vascular cell adhesion molecule (VCAM) and intercellular adhesion molecule (ICAM)
Endo-peripheral artery tonometry (EndoPAT) index | 6 weeks
  EndoPAT index was assessed to evaluate endothelial function by using a finger plethysmograph based on non-invasive peripheral artery tonometry.

CONTACTS AND LOCATIONS:
Overall Officials: Nan Hee Kim, Prof, Principal Investigator — Department of Endocrinology and Metabolism, Korea University Ansan Hospital
Locations (1):
- Department of Endocrinology and Metabolism, Korea University Ansan Hospital, Ansan-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Lee YJ, Seo JA, Yoon T, Seo I, Lee JH, Im D, Lee JH, Bahn KN, Ham HS, Jeong SA, Kang TS, Ahn JH, Kim DH, Nam GE, Kim NH. Effects of low-fat milk consumption on metabolic and atherogenic biomarkers in Korean adults with the metabolic syndrome: a randomised controlled trial. J Hum Nutr Diet. 2016 Aug;29(4):477-86. doi: 10.1111/jhn.12349. Epub 2016 Mar 6. PMID 26945812